



| For participation in:* | Behavioural | EEG | Sled | Robot |
|------------------------|-------------|-----|-----------|--------------------|
| | | | *tick the | applicable box(es) |

## To be filled out by the PARTICIPANT:

- I was satisfactorily informed about the study both verbally and in writing, by means of the general information brochure (version 3.0) and additional study specific information brochure(s).
- I was able to ask questions about the study which have been answered adequately. I had enough time to decide if I want to take part.
- I know that taking part in the study is voluntary. I also know that I can decide not to take part or stop taking part at any moment. I do not have to explain why.
- I give consent to the researchers to collect and use my research data for a minimum period of 10 years.
- I give consent to acquisition of personal data for administrative purposes.
- I give consent to collect demographic data (like gender or age) to answer the research question.

## I understand that:

- I have the right to withdraw from the experiment at any time without having to give a reason.
- My research data are not examined from a clinical perspective.
- I have the right to request disposal of my research data that are potentially identifiable up to 1 month after finalization of the data collection.

PLEASE TURN OVER THIS PAGE

## Please tick yes or no in the below table and include the date.

| I give my consent to participate in this experiment. | | No* |
|---|---|---|
| I give my consent that sensitive personal data on my health, background or | | No* |
| preferences is collected to answer the research question. | | |
| For reviewing purposes some authorities will be able to see all of my data. | Yes | No* |
| These authorities are mentioned in the information brochure. I give consent | | |
| to these to access and review my data. | | |
| I give my consent that my not directly identifiable experimental data will be | Yes | No* |
| collected and stored. | | |
| I give my consent that my not directly identifiable experimental data will be | Yes | No* |
| made public, e.g. the data are publicly shared with persons interested in the | | |
| data, for instance for verification, re-use and/or replication. | | |
| Datum | | // |
| data, for instance for verification, re-use and/or replication. | | _ |

\*If you answer one of the questions above with 'no', then you cannot participate in this experiment.

| I give consent to approach me after this study to participate in a follow-up study and understand that the coupling between my personal contact details and the research data is stored. At the latest this is deleted one month after finalization of the research. | Yes | No** |
|---|---|---|
| I give my consent that some sensitive personal data on my health, background or preferences is made public, e.g. the data are publicly shared with persons world-wide who are interested in the data, for instance for verification, re-use and/or replication. | Yes | No** |

<sup>\*\*</sup>The answer to these questions does not affect participation in this research. Hence you can answer with 'no' and still participate.

| To be filled out by the RESEARCHER prior to the start of the I declare that I have provided this participant with all the information | ne experiment: | | | |
|---|---|---|---|---|
| Name researcher (or the representant of the researcher: | | | | <br> |
| PI group: | | | | <br> |
| DCC PPF number: | | | | <br> |
| Participant number | | | | <br> |
| Signature: | Date: | 1 | 1 | |